CLINICAL TRIAL: NCT01075230
Title: A Prospective, Randomized, Single-blind, Multi-center Clinical Study to Evaluate the Effect of Platelet Rich Plasma (PRP) on Short-term Patient Outcomes Following Total Knee Replacement.
Brief Title: Standard Total Knee Arthroplasty Using Platelet Rich Plasma (PRP)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intended as multi-center. 1 of 2 sites could not participate. Enrollment discontinued after 50/100. Subjects followed per protocol.
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR08-004
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis
Keywords: PRP, TKA, pain scale, hemoglobin, hematocrit, narcotics
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard TKA (Active Comparator): Subjects in this arm will receive total knee replacement as standard of care without Platte Rich Plasma
  Interventions: Procedure: Total knee arthroplasty
- Standard TKA with PRP (Active Comparator): Subjects in this arm will receive total knee replacement as standard of care with Platte Rich Plasma
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Subject will undergo total knee arthroplasty according to established surgeon / hospital protocol.
  Other Names: Optetrak total knee system

SUMMARY:
Clinical study to determine if there is a difference in hemoglobin level between patients undergoing total knee arthroplasty with and without platelet-rich plasma.

DETAILED DESCRIPTION:
The purpose of this study is to determine if there is a difference in hemoglobin level between patients undergoing total knee arthroplasty with and without platelet-rich plasma.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female who is undergoing primary unilateral surgery or the first surgery of a staged bilateral total knee replacement where the second stage will be at least 6 weeks later
* Patient agrees to be blinded to their treatment group assignment
* Patient is willing and able to return for follow-up over at least a six (6) month post-operative period although longer follow-up may be desired
* Patient agrees to participate by signing an IRB approved Informed Consent Form

Exclusion Criteria:

* Patient will have a staged bilateral total knee replacement with the second stage to be performed less than 6 weeks after the first stage surgery PRP in
* Patient has had previous surgery on the operative knee that will necessitate the removal of existing hardware (e.g. previous osteotomy)
* Patient has a known adverse reaction or sensitivity to bovine (cow) thrombin (used as part of the platelet rich plasma system) or other bovine-derived products
* Patient has hemoglobin < 12.0 (males), < 11.0 (females)
* Patient has a clinically significant anxiety disorder
* Patient is on therapeutic anticoagulation medication and has an INR > 1.3
* Patient has a severe bleeding disorder
* Patient has a known addiction to drugs or alcohol, including, but not limited to: chronic daily use of narcotic medications for more than 90 days prior to surgery
* Patient is pregnant
* Patient is a prisoner
* Patient is involved in a personal litigation (e.g. Worker's Compensation) that relates to their knee surgery
* Patient is actively participating in another medical device, drug, or biologic clinical trial (active defined as having treatment within the last 30 days)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin (Hgb) level | Preop, post-op day 2
  Hemoglobin level analysis

SECONDARY OUTCOMES:
Visual analog scale (VAS) for pain | Preop, post-op day 1, post-op day 2, discharge, 6 weeks
  Visual analog scale for Pain (1-10), 10 being the worst

CONTACTS AND LOCATIONS:
Locations (1):
- Henrico Doctors' Hospital, Richmond, Virginia, United States